CLINICAL TRIAL: NCT04548674
Title: Effect of Different Desensitizing Protocols on the Pulp Inflammatory Response in Bleached Teeth: A Randomized Clinical Trial.
Brief Title: Analysis of the Influence of Desensitizing Treatments on the Pulp Inflammatory Response in Bleached Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Para (Other)
Responsible Party: Principal Investigator, Cecy Martins Silva, Professor Clínico, Universidade Federal do Para
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: UFPara-008
Record Dates: First submitted 2020-09-01; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Pulp Inflammation
Keywords: Therapies; Caspase 3; Immunohistochemistry
MeSH Terms: conditions — Spinocerebellar Ataxias | interventions — Lasers; 6-chloro-2-(1-piperazinyl)pyrazine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Positive Control Group (Placebo Comparator): Whiteness HP 35%
  Interventions: Other: Whiteness HP 35%
- Laser Group (Experimental): Whiteness HP 35% + Laser
  Interventions: Other: Whiteness HP 35%; Device: Whiteness HP 35% + LASER
- CPP Group (Experimental): Whiteness HP 35% + CPP
  Interventions: Other: Whiteness HP 35%; Other: Whiteness HP 35% + CPP
- Nano Group (Experimental): Whiteness HP 35% + NANO
  Interventions: Other: Whiteness HP 35%; Other: Whiteness HP 35% + NANO
- Negative Control (No Intervention): Without intervention

INTERVENTIONS:
Other: Whiteness HP 35% — Single application of 45 minutes on the buccal surfaces of third molars, with an average thickness of 1 mm
  Arms: CPP Group; Laser Group; Nano Group; Positive Control Group
Device: Whiteness HP 35% + LASER — A dose of LASER (60 J / cm2, for 16 seconds) was applied at two points, one point in the cervical region and another in the center of the buccal surface of the third molars, using visible infrared LASER therapy (Photon III / DMC, São Carlos, SP, Brazil), with a wavelength of 808 nm, and AsGaAl, as an active medium.
  Arms: Laser Group
Other: Whiteness HP 35% + CPP — Topical application of casein phosphopeptide amorphous calcium phosphate fluoride CPP-ACPF (My Paste Plus, Recaldent, GC, USA) with the aid of a microbrush (KG Sorensen, SP, Brazil) in a passive way for 5 minutes.
  Arms: CPP Group
Other: Whiteness HP 35% + NANO — A topical application of nanohydroxyapatite (Nano P FGM, SC, Brazil) was performed with the aid of a microbrush (KG Sorensen, SP, Brazil) in a passive way for 5 minutes after teeth whitening.
  Arms: Nano Group

SUMMARY:
This randomized, controlled, blinded clinical trial evaluated the effectiveness of different desensitizing protocols in preventing pulp inflammation after bleaching treatment with 35% hydrogen peroxide (PH) (Whiteness PH 35%).

DETAILED DESCRIPTION:
Thirty healthy third human molars extracted by orthodontic indication were randomized and allocated into five groups (n = 6): CN (negative control): without intervention; CP (Positive control): PH; PMB: PH + photobiomodulation with low power laser; CPP: PH + casein phosphopeptide phosphopeptide amorphous calcium phosphate (CPP-ACPF); NANO: PH + nanohydroxyapatite. The office whitening was performed in two sessions with a single application of 45 min and an interval of 48 hours between them. Pulp tissues were removed for immunohistochemical analysis. Immunostaining was performed for Caspase 3 using an Axio Scope.A1 microscope.

ELIGIBILITY:
Inclusion criteria:

* Lower third molars class I position A
* Maxillary third molars horizontal position A
* Absence of caries and enamel fracture
* Absence of periodontal disease
* Extraction of third molars for orthodontic reasons
* No allergy to the anesthetic and positive pulp sensitivity test

Exclusion criteria:

* Calcification in the middle third of the root
* Drug users or smokers
* Patients who have already done whitening
* Root apex with incomplete formation and patients with systemic problems that would make surgery impossible

Ages: 20 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Pulp inflammation | 3 days After extraction of third molars
  Evaluation of pulp inflammation through immunohistochemistry of the third molar whitening or not

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal do Pará, Belém, Pará, Brazil